CLINICAL TRIAL: NCT00113243
Title: Phase I Study of Stem Cell Mediated Angiogenesis for Limb Threatening Ischemia
Brief Title: Safety Study of Using Stem Cells to Stimulate Development of New Blood Vessels in Peripheral Vascular Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Murphy, Michael P., MD (Individual)
Collaborators: Indiana University School of Medicine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUPUI 0503-14
Record Dates: First submitted 2005-06-06; First posted 2005-06-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

INTERVENTIONS:
Drug: adult stem cells

SUMMARY:
The purpose of this study is to determine if bone marrow derived adult stem cells are safe and effective in inducing development of new blood vessels (angiogenesis) in the legs of patients with severe peripheral vascular disease.

DETAILED DESCRIPTION:
Presently there are no effective medical therapies to enhance blood flow in the legs of patients with peripheral vascular disease. For patients with limb threatening ischemia the only option for relief of rest pain or gangrene is amputation.

There is evidence in animal and clinical studies that adult stem cells in the bone marrow, called endothelial progenitor cells, participate in the development of new blood vessels, a process called angiogenesis. In this investigation, patients with limb threatening ischemia will have their bone marrow harvested and the stem cells will then be removed and injected directly into the muscle of the diseased leg. The procedure will require about 4 hours and the subjects will be admitted to the Indiana University Medical Center overnight. The follow-up period is 12 weeks and the analysis will consist of examinations at 1, 2, 4, 6, 8, and 12 weeks. Adverse and serious adverse events will be recorded during this time period. Diagnostic studies will be obtained to measure blood flow in the treated leg during the follow up period and include transcutaneous (skin) oxygen measurements, pressure recordings in the leg, arteriography, magnetic resonance imaging, and wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Severe peripheral vascular disease not amenable to bypass or angioplasty
* Age >21 years old
* Normal renal function (creatinine < 1.6)

Exclusion Criteria:

* Congestive heart failure (ejection fraction [EF]<30%)
* History of cancer or myeloproliferative disorders
* Proliferative retinopathy
* Pregnancy
* Cognitively disabled

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-12; Study Completion 2007-12

PRIMARY OUTCOMES:
Adverse events recorded in the 12 week study period
Serious Adverse events recorded for one year

SECONDARY OUTCOMES:
Changes in limb perfusion after treatment with stem cells will be assessed with arteriography, blood pressure recordings, oxygen measurements, and wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Murphy, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Rehman J, Li J, Parvathaneni L, Karlsson G, Panchal VR, Temm CJ, Mahenthiran J, March KL. Exercise acutely increases circulating endothelial progenitor cells and monocyte-/macrophage-derived angiogenic cells. J Am Coll Cardiol. 2004 Jun 16;43(12):2314-8. doi: 10.1016/j.jacc.2004.02.049. PMID 15193699
- [Background] March KL, Johnstone BH. Cellular approaches to tissue repair in cardiovascular disease: the more we know, the more there is to learn. Am J Physiol Heart Circ Physiol. 2004 Aug;287(2):H458-63. doi: 10.1152/ajpheart.00343.2004. No abstract available. PMID 15277189
- [Background] Rehman J, Li J, Orschell CM, March KL. Peripheral blood "endothelial progenitor cells" are derived from monocyte/macrophages and secrete angiogenic growth factors. Circulation. 2003 Mar 4;107(8):1164-9. doi: 10.1161/01.cir.0000058702.69484.a0. PMID 12615796
- [Derived] Liang TW, Jester A, Motaganahalli RL, Wilson MG, G'Sell P, Akingba GA, Fajardo A, Murphy MP. Autologous bone marrow mononuclear cell therapy for critical limb ischemia is effective and durable. J Vasc Surg. 2016 Jun;63(6):1541-5. doi: 10.1016/j.jvs.2016.01.022. Epub 2016 Mar 23. PMID 27021379
- See also: General Clinical Research Center at Indiana University School of Medicine — http://www.gcrc.iupui.edu/